CLINICAL TRIAL: NCT05367947
Title: Investigation of In-phase Bilateral Exercise Effects on Corticospinal Plasticity in Relapsing Remitting Multiple Sclerosis: a Registered Report Single-case Concurrent Multiple Baseline Design Across Five Subjects
Brief Title: In-phase Bilateral Exercises in People With Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: The Cyprus Foundation for Muscular Dystrophy Research (Other)
Responsible Party: Principal Investigator, Dimitris Sokratous, Mr, Cyprus University of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IBEMS
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: transcranial magnetic stimulation; multiple sclerosis; exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study follows a concurrent multiple baseline design across subjects, which involves five people with RRMS that will be managed as five different case studies. The specific design has the advantage to verify the cause-effect inference clearly by the staggered duration through separate baseline phases
Masking Description: Participants are people with multiple sclerosis according inclusion/exclusion criteria.
  Investigators are health professionals (i.e., physiotherapist, sports scientist, neuropsychologist, neurologist, biostastician).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-phase bilateral RRMS Participants A-E (Experimental): The study follows a concurrent multiple baseline design across subjects, which involves five people with RRMS as five different case studies.
  Interventions: Behavioral: In-phase Bilateral Exercises of the upper limbs

INTERVENTIONS:
Behavioral: In-phase Bilateral Exercises of the upper limbs — The intervention protocol consists of in-phase bilateral exercises for the upper limbs, which are adapted to different sport activities and to fitness functional exercises, organized in a circuit training. Specifically, each session will consist of 1-3 sets, consisting of 10-15 repetitions of 9 different exercises targeting large muscle groups of the upper limbs.
  The specific exercises will include sports activities of basic technical skills of basketball (e.g., different types of passing, catching and throwing the ball) and volleyball (e.g., different types of passing and receiving the ball), whereas the fitness exercises will include shoulder rows, shoulder lateral raises, elbow flexions, elbow extensions, using resistance elastic bands, as well as exercises with the patients' own body weight (e.g., pushups, TRX).
  The intervention phase for each participant will consist of 12 consecutive weeks, for 3 times per week, 30-60 minutes each session.

SUMMARY:
Relapsing-remitting multiple sclerosis (RRMS) is associated with changes of the corticospinal tract integrity, which is quantified by means of corticospinal plasticity. Several factors, such as exercise and interlimb coordination can influence such corticospinal plasticity. Previous work in healthy and in stroke participants showed that the greatest improvement of corticospinal plasticity occurred during in-phase bilateral arm exercises. Here, the investigators propose a concurrent multiple baseline design study which has the advantage to verify the cause-effect inference by the staggered duration through separate baseline phases. The proposed study includes five people with RRMS, who will follow an intervention protocol which includes in-phase bilateral movements of the upper limbs, adapted to different sports activities and to functional training. The aim of the study is to investigate the effects of in-phase bilateral exercises on corticospinal plasticity and on clinical measures, using transcranial magnetic stimulation and standardized clinical assessment. To meet quality standards, the present study has been designed and will be conducted according to the "What Works Clearinghouse" criteria for single case studies.

DETAILED DESCRIPTION:
Relapsing-remitting multiple sclerosis (RRMS) is the most common type of multiple sclerosis characterized by periods of relapses and generating various motor symptoms. These symptoms are associated with the corticospinal tract integrity neuroplasticity. The corticospinal tract is one of the major motor descending pathways providing voluntary motor function in humans. The neuroplasticity of the corticospinal tract, as defined by changes in neuron structure or function detected either directly from measures of individual neurons or inferred from measures taken across populations of neurons, is an essential factor that predicts clinical recovery in the post-relapse stage of people with RRMS. Corticospinal plasticity can be probed using Transcranial Magnetic Stimulation (TMS) and characterized via certain TMS-specific neurophysiological measures. Corticospinal plasticity is exercise-dependent and influenced by various factors, such as aerobic exercise, resistance training, as well as interlimb coordination. Previous studies that assessed corticospinal plasticity using TMS in healthy participants and in chronic stroke survivors, reported that interlimb coordination and especially in-phase bilateral movement has the strongest effect on corticospinal plasticity.

Despite the broad literature on the effects of different types of exercises on the neuroplasticity in people with RRMS, it is unclear whether in-phase bilateral exercises can promote motor related neuroplastic changes in RRMS. In light of evidence that people with RRMS have bilateral cortical lesions, which cause bilateral changes of corticospinal tract integrity, these findings raise the question about the effects of in-phase bilateral exercises on corticospinal plasticity. Such effects would provide strong evidence about whether exercise, in particular in-phase bilateral exercise, can influence the corticospinal plasticity in RRMS.

The aim of this concurrent multiple baseline design study is to investigate the effects of in-phase bilateral exercises on corticospinal plasticity and on clinical measures using TMS and standardized clinical assessment, in five people with RRMS. The intervention protocol will last for 12 consecutive weeks (30-60 minutes /session x 3 sessions/week) and include in-phase bilateral movements of the upper limbs, adapted to different sports activities and to functional training.

To define functional relation between the intervention and the results on corticospinal plasticity (i.e., resting motor threshold, motor evoked potential amplitude, latency) and on clinical measures (i.e., balance, gait, bilateral hand dexterity and strength, cognitive function), the investigators will perform a visual analysis followed by multilevel modelling and the single case educational design specific mean difference in order to estimate the magnitude of the effect size across cases.

Visual analysis will conducted first, in order to determine whether there is a functional relationship between the intervention and the outcome measures. During the visual analysis, six features of the research design graphed data will be examined: level, trend, stability, immediacy of the effect, overlap, and consistency. Over the within-phase examination an evaluation of level, trend and stability will be examined. Level will be reported from the mean score of each dependent variable and trend will determine whether the data points are monotonically decreased or increased. Stability will be estimated based on the percentage of data points falling within 15% of the phase median, if this is higher than 80% then we assume that this criterion is met. Additionally, over the between-phase examination an evaluation of overlapping data among baseline and intervention phases, consistency of data patterns and immediacy of effect will be performed. The Percentage of Non-overlapping Data index will be used to quantify the proportion of data points in the intervention phase that do not overlap with the baseline phase and the test statistic will be calculated using the Improvement Rate Difference as an effect size index. Immediacy of the effect will be examined by comparing changes in level between the last three data points of one phase and the three first data points of the next phase. Furthermore, consistency of data patterns involves the observation of the data from all phases within the same condition, with greater consistency expressing greater causal relation. Each feature will be assessed individually and collectively across to all participants and to all phases. Consequently, if the intervention protocol is the sole determinant of improvement, the investigators expect to find indicators of improvement only at the intervention phase.

Secondly, a quantitative analysis methods will conducted so to evaluate the magnitude of the intervention effect, provided there is evidence from the visual analysis. The investigators will perform all neurophysiological and clinical assessments to each participant according to the number of data points during each phase (i.e., baseline, intervention, follow up). In order to estimate the individual-level effect sizes, three different methods will be used, as suggested by 'What Works Clearinghouse', the standardized mean difference (Cohen's d), the standardized mean difference with correction for small sample sizes (Hedges' g) and piecewise regression analysis which does not only reflect the immediate intervention effect, but also the intervention effect across time. Multilevel modelling, which is recommended by the 'What Works Clearinghouse' and the single case educational design, specific mean difference index will be used to estimate the magnitude of the effect across cases and compared to the effect obtained by the single level estimates. All tests will be two sided. Statistical analysis will be performed using the statistical software R (https://www.r-project.org/).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with relapsing remitting multiple sclerosis
* Expanded Disability Status Scale score between three and five
* Aged between 30 and 70 years
* Relapse within 30 days
* Mini Mental State of Examination score between 24 and 30 (no cognitive impairment)

Exclusion Criteria:

* Metal implants
* History of any disease affecting the central nervous system other than multiple sclerosis
* History of cardiovascular disease
* Mental disorders
* Severe orthopedic disorders
* Pregnancy
* Visual deficit
* Hearing impairments,
* Εpileptic seizures
* Spasticity level on upper or lower limbs more than 1+ (slight increase in muscle tone) according to Modified Ashworth Scale

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Corticospinal Plasticity | Through study completion, an average 35 weeks
  The investigators will assess the corticospinal plasticity using single pulse Transcranial Magnetic Stimulation (TMS). Following TMS recommended guidelines concerning safety and experimental conditions, bilateral cortical excitability and bilateral central motor conduction time (CMCT) will be assessed. Using electromyography (EMG) signals, the investigators will analyze bilateral cortical excitability and bilateral CMCT to determine corticospinal plasticity. The resting motor threshold (rMT) and the Motor Evoked Potential (MEP) amplitude of Abductor Pollicis Brevis muscle will define cortical excitability, while the MEP latency will be used to calculate the CMCT. To ensure methodological consistency, the investigators will collect all data by performing the same methodological procedures for both conditions (i.e., cortical excitability and CMCT) bilaterally (one side per assessment), across participants and across all time points.

SECONDARY OUTCOMES:
Mini Balance Evaluation Systems Test | Through study completion, an average 35 weeks
  It measures dynamic balance, functional mobility, and gait in neurological patients, including people with multiple sclerosis. The specific test consists of 14 items, including four of the six segments (anticipatory postural adjustments, sensory orientation, reactive postural control and dynamic gait) from the Balance Evaluation Systems Test.
Six Spot Step Test | Through study completion, an average 35 weeks
  It is a timed walking test that involves kicking over a number of targets placed along a 5m-path in which rely to some extent on vision and cognition. The Six Spot Step Test is measured in the time domain replicating a complex range of sensorimotor functions, part of which are lower limb strength, spasticity, coordination, as well as balance
Action Research Arm Test | Through study completion, an average 35 weeks
  It is a 19-item observational measure used by physiotherapists and other health care professionals to examine upper limb performance (i.e., coordination, dexterity and functioning). Items covering the Action Research Arm Test are categorized into four subscales (grasp, grip, pinch and gross movement).
Isometric Dynamometer | Through study completion, an average 35 weeks
  We well assess the isometric muscle force of major muscle groups with the use of a hand held dynamometer, which is used in the evaluation and rehabilitation of muscle strength. Shoulder flexors, extensors, rotators, horizontal adductors and abductors adductors and abductors, elbow flexors and extensors are the major muscle groups which will be evaluated.
Symbol Digit Modalities Test | Through study completion, an average 35 weeks
  We will employ the oral form which assesses the information processing speed. During the test, the participant will be given two minutes to orally match symbols with digits as quickly as possible.
Modified Fatigue Impact Scale | Through study completion, an average 35 weeks
  It is a short questionnaire which requires the participants to describe the effects of fatigue during the past four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Sokratous, MS, Study Director — Cyprus University of Technology
Locations (1):
- Dimitris Sokratous, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Neva JL, Lakhani B, Brown KE, Wadden KP, Mang CS, Ledwell NH, Borich MR, Vavasour IM, Laule C, Traboulsee AL, MacKay AL, Boyd LA. Multiple measures of corticospinal excitability are associated with clinical features of multiple sclerosis. Behav Brain Res. 2016 Jan 15;297:187-95. doi: 10.1016/j.bbr.2015.10.015. Epub 2015 Oct 20. PMID 26467603
- [Background] Pascual-Leone A, Tarazona F, Keenan J, Tormos JM, Hamilton R, Catala MD. Transcranial magnetic stimulation and neuroplasticity. Neuropsychologia. 1999 Feb;37(2):207-17. doi: 10.1016/s0028-3932(98)00095-5. PMID 10080378
- [Background] Whitall J, Waller SM, Sorkin JD, Forrester LW, Macko RF, Hanley DF, Goldberg AP, Luft A. Bilateral and unilateral arm training improve motor function through differing neuroplastic mechanisms: a single-blinded randomized controlled trial. Neurorehabil Neural Repair. 2011 Feb;25(2):118-29. doi: 10.1177/1545968310380685. Epub 2010 Oct 7. PMID 20930212
- [Background] Smith AL, Staines WR. Cortical and behavioral adaptations in response to short-term inphase versus antiphase bimanual movement training. Exp Brain Res. 2010 Sep;205(4):465-77. doi: 10.1007/s00221-010-2381-5. Epub 2010 Aug 14. PMID 20711566
- [Background] Neva JL, Legon W, Staines WR. Primary motor cortex excitability is modulated with bimanual training. Neurosci Lett. 2012 Apr 18;514(2):147-51. doi: 10.1016/j.neulet.2012.02.075. Epub 2012 Mar 3. PMID 22405809
- [Background] Kratochwill, T. R. Hitchcock, J. Horner, R. H. Levin, J. R. Odom, S. L. Rindskopf, D. M Shadish WR. Single-Case Design Technical Documentation. Work Clear website http//ies.ed.gov/ncee/wwc/pdf/wwc_scd.pdf. 2010;(December):2010.
- [Background] Zhan S, Ottenbacher KJ. Single subject research designs for disability research. Disabil Rehabil. 2001 Jan 15;23(1):1-8. doi: 10.1080/09638280150211202. PMID 11213316
- [Background] Lobo MA, Moeyaert M, Baraldi Cunha A, Babik I. Single-Case Design, Analysis, and Quality Assessment for Intervention Research. J Neurol Phys Ther. 2017 Jul;41(3):187-197. doi: 10.1097/NPT.0000000000000187. PMID 28628553
- [Derived] Sokratous D, Charalambous CC, Zamba-Papanicolaou E, Michailidou K, Konstantinou N. A 12-week in-phase bilateral upper limb exercise protocol promoted neuroplastic and clinical changes in people with relapsing remitting multiple sclerosis: A registered report randomized single-case concurrent multiple baseline study. PLoS One. 2024 Oct 17;19(10):e0299611. doi: 10.1371/journal.pone.0299611. eCollection 2024. PMID 39418242
- [Derived] Sokratous D, Charalambous CC, Papanicolaou EZ, Michailidou K, Konstantinou N. Investigation of in-phase bilateral exercise effects on corticospinal plasticity in relapsing remitting multiple sclerosis: A registered report single-case concurrent multiple baseline design across five subjects. PLoS One. 2023 Mar 2;18(3):e0272114. doi: 10.1371/journal.pone.0272114. eCollection 2023. PMID 36862693